CLINICAL TRIAL: NCT05137977
Title: Is Invasive ICU-treatment Associated With Mental Illness?
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: RBM2021
Record Dates: First submitted 2021-11-16; First posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Postintensive Care Syndrome; Anxiety Disorder; Depression; PTSD; PICS; Intensive Care Psychiatric Disorder
MeSH Terms: conditions — postintensive care syndrome; Anxiety Disorders; Depression; Stress Disorders, Post-Traumatic | interventions — Critical Care; Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SIR: All adult intensive care patients. Data from the The Swedish intensive care registry
  Interventions: Procedure: Intensive Care

INTERVENTIONS:
Procedure: Intensive Care — Invasive ventilation more than 24hs.
  Other Names: CRRT; Invasive ventilation

SUMMARY:
Understanding long-term complications after intensive care is important to be able to offer prophylactic and therapeutic measures to post-intensive care unit (ICU) patients.

Since patients in the ICU experience life threatening conditions, severe psychological and physical stress, we hypothesized that patients after ICU have an increased risk of mental illnesses specifically anxiety disorders, depression and post-traumatic stress disorder (PTSD). Moreover, we hypothesized that the prevalence and severity of mental illnesses are related to the extent of intensive care.

Our endpoints are the prevalence of anxiety disorders, depression one year after ICU-care and if the extent of intensive care an independent predictor of psychiatric illness one year after ICU admission.

We will assess Swedish Intensive Care registry data for all adult ICU patients admitted between 2010-2015 and assess ICD-10 codes for anxiety disorders, depression and PTSD one year after ICU admission.

DETAILED DESCRIPTION:
Background

As intensive care unit (ICU)-mortality rates are improving in many areas, research focus has turned towards sequelae after ICU-care. The term Post Intensive Care Syndrome has been coined, concluding a high frequency of mental illness, cognitive and physical impairment immediately after ICU-care. Since patients in the ICU experience life threatening conditions, severe psychological and physical stress, we hypothesize that patients after ICU have an increased risk of long-term mental illnesses that increase with the extent of intensive care, specifically anxiety, and post-traumatic stress disorder (PTSD). Current data on the extent and severity of mental illness after intensive care, and if intensive care is an independent predictor of it, is limited.

Objective

Our objective is to assess in nationwide data if extensive ICU-treatment contributes to mental illness. Extensive ICU-treatment will be defined in our dataset as ICU-treatment of patients in need of invasive ventilation, and/or continuous renal replacement therapy (CRRT). Our endpoints are prevalence of mental illness one year after discharge, and its association between extent of ICU-treatment.

Method

We will use the Swedish intensive Care registry of intensive care patients treated between 2010 and 2015 for extracting data on Data on Invasive ventilation treatment, CRRT-treatment, gender and age. ICD-10 codes corresponding for anxiety, PTSD and depression, and other diagnoses known to increase the risk of mental illness will be extracted from the Swedish National Patient Registry. Patients younger than 18 years old and ICU-codes corresponding for pre-existing anxiety, PTSD, depression, and treatment periods less than 24 hours will be excluded from the study. Missing data will be imputed. A multivariable regression model will be fit using ICU-codes corresponding with mental illness as dependent variable, Invasive ventilation and CRRT as independent variables, and the other parameters as covariates.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old

Exclusion Criteria:

* ICD codes for previous mental illness.
* ICU stay less than 24 hours

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Nationwide registry of patients admitted to ICU treatment in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 1048576 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Mental illness | 2010-2015
  Defined as PTSD, depressive symptoms or anxiety or combination of the earlier mentioned.